CLINICAL TRIAL: NCT01166802
Title: Development of a Questionnaire to Measure Hypervigilance for Visceral Pain
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: William E Whitehead, PhD/Professor of Medicine, University of North Carolina, Chapel Hill
Other Study IDs: 07-005L
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: questionnaire development; hypervigilance; pain sensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to develop and validate a questionnaire (non-invasive technique) to identify patients who are hypervigilant for noxious visceral sensations and who show a lower threshold to report pain. This questionnaire would be useful in studies investigating the role of visceral pain hypervigilance and pain sensitivity in the comorbidity of IBS with other somatic disorders.

DETAILED DESCRIPTION:
Methods: There are two phases to the project: (1) Development of the pool of items (questions), and (2) validating individual items based on their correlation with an objective gold standard - the response criterion statistic, B, calculated from a barostat test of pain sensitivity. We will perform barostat tests of pain thresholds and other measures of pain sensitivity that are based on sensory decision theory analysis in a relatively large group of 84 IBS patients. Sensory decision theory divides pain perception into two components: a perceptual sensitivity index (P(A)) and a response criterion (B). The response criterion is sensitive to cognitive and psychological influences on pain perception. We will use this index (B) as the gold standard against which to select items for a scale to measure hypervigilance for visceral pain. The process will involve (a) pooling items from existing questionnaires that seem related to the concept, (b) obtaining additional questions from consultants who are experts in visceral perception and psychometric test development, (c) identifying the items that show the strongest correlations with the response criterion, (d using principal components analysis to reduce the items to the smallest number of non-redundant items that predict the response criterion and treating this as a provisional questionnaire of hypervigilance, and (e calculating psychometric characteristics of this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of IBS
* meets Rome III criteria for IBS
* women or men aged 18 or older

Exclusion Criteria:

* use of IBS-specific compounds, opiates, anticholinergics, or any drug likely to cause constipation as a side-effect
* use of analgesics for 48 hours prior to the study
* hypothyroid
* history of bowel resection except appendectomy or cholecystectomy
* psychotic disorder, major depression, substance abuse (other than tobacco)or other psychiatric condition likely to interfere with the conduct of the study
* renal disease
* patients with inflammatory or ischemic disease of the rectum
* known to be unreliable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with irritable bowel syndrome, age 18 or older, of any race or gender, will be enrolled. These subjects will be recruited from the Functional GI & Motility Disorder's Registry of Research Participants.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center for Clinical and Translational Research, Chapel Hill, North Carolina, United States